CLINICAL TRIAL: NCT04771013
Title: A Single-arm, Open-Label, Phase II Clinical Study to Evaluate the Safety and Efficacy of Thymic Peptides in the Treatment of Hospitalized COVID-19 Patients in Honduras
Brief Title: Safety and Efficacy of Thymic Peptides in the Treatment of Hospitalized COVID-19 Patients in Honduras
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Católica de Honduras (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Héctor Miguel Ramos Zaldívar, Director of the Catholic University of Honduras Medical Research Group (GIMUNICAH), Universidad Católica de Honduras
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEC-01-2021; COM-2020-01 (Other: Catholic University of Honduras IRB in Tegucigalpa); AEC-01-2021 (Registry Identifier: Dirección General de Vigilancia del Marco Normativo Honduras)
Record Dates: First submitted 2021-02-24; First posted 2021-02-25 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 Infection; COVID-19 Pandemic; 2019 Novel Coronavirus Disease; Thymic peptides; Thymus gland; Peptides; Honduras; Coronavirus Disease 2019; Coronavirus Disease-19; COVID-19 Virus Infection; 2019-nCoV Disease; 2019-nCoV Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A participant-level comparison based on registry data from the Hospital de Santa Bárbara Integrado will be performed after propensity score matching.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daily oral dose of thymic peptides (Experimental): Patients will receive a daily oral dose of 250 mg of lyophilized thymic peptides dissolved in 50 mL of water (one hour before or two hours after a meal) in addition to the standard treatment, for up to 20 days or until medical discharge.
  Interventions: Biological: Thymic peptides

INTERVENTIONS:
Biological: Thymic peptides — 250 mg oral daily dose of lyophilized thymic peptides dissolved in 50 mL of water, administered with an empty stomach.
  Other Names: Unicahsina

SUMMARY:
This is a single-arm, open-label, phase II clinical study to evaluate the safety and efficacy of thymic peptides in the treatment of hospitalized COVID-19 patients in Honduras.

DETAILED DESCRIPTION:
This study was approved and registered by the Dirección General de Vigilancia del Marco Normativo de la Secretaría de Salud de Honduras (General Directorate for Regulatory Framework Surveillance of the Ministry of Health of Honduras) the eight of February of 2021; enrollment began tenth of February of 2021.

The study will analyze 23 clinical parameters, 9 laboratory studies besides complete blood count, chest radiography, time to response, adverse clinical outcomes, and hospital length of stay in 22 participants treated with a daily oral dose of 250 mg of lyophilized thymic peptides dissolved in 50 mL of water (one hour before or two hours after a meal) in addition to the standard treatment. A participant-level comparison based on registry data from Hospital de Santa Bárbara Integrado will be performed after propensity score matching. The Generic Assessment of Side Effects in Clinical Trials (GASE) will be applied in addition to monitoring of treatment-emergent adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed case of COVID-19 by viral nucleic acid (RNA) detection, viral antigen detection, or detection of antibodies to the virus.
* Participants that require hospitalization under Honduran Ministry of Health Guidelines for Clinical Management of COVID-19 Adult Patients: Stage IIb, defined as a patient with or without risk factors that presents with warning signs (shortness of breath, tachypnea), and altered inflammatory parameters.
* Participants that present with at least one of the following: oxygen saturation level below 94 percent; complete blood count showing lymphopenia, neutrophilia, or both; positive C-reactive protein; chest radiography or CT scan with ground-glass opacities.
* Male or female at least 21 years old.

Exclusion Criteria:

* COVID-19 patients that do not require hospitalization under Honduran Ministry of Health Guidelines for Clinical Management of COVID-19 Adult Patients: phase IA (asymptomatic), phase IB (mild symptoms without risk factors), or phase IC (mild symptoms with risk factors).
* Participants currently in other clinical trials evaluating experimental drugs.
* Known history of allergic reactions to thymic peptides or calf thymus acid lysate derivatives.
* Organ transplant recipients.
* Women who are pregnant or breast feeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Héctor M Ramos, MD, Study Director — Universidad Católica de Honduras; Pontificia Universidad Católica de Chile; Karla G Reyes, MD, Principal Investigator — Universidad Católica de Honduras; Universidad Mayor; Nelson A Espinoza, MD, Principal Investigator — Universidad Católica de Honduras
Locations (1):
- Hospital de Santa Bárbara Integrado, Santa Bárbara, Honduras

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For individual participant data meta-analysis.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 participants were enrolled in the intervention group.
  A participant-level comparison based on a control group by propensity score matching from registry data was performed. This accounts for the 22 patients in the arm of the historic control group.
  ClinicalTrials.gov Identifier: NCT04771013
  MedRxiv: A nonrandomized phase 2 trial of oral thymic peptides in hospitalized patients with Covid-19. doi: https://doi.org/10.1101/2021.12.05.21267318
Groups:
- Historic Control Group: A participant-level comparison based on a control group by propensity score matching from registry data was performed.
  For the comparison group, registry data from June 2020 to February 2021 was considered, as standardization of Stage IIB therapeutic management to its current guideline in Honduras occurred on May 2020.
  Although highly controversial among the Honduran scientific community, guidelines approved by the Honduran Ministry of Health for the treatment of Covid-19 include the use of ivermectin, azithromycin, zinc, hydroxychloroquine or chloroquine, acetaminophen, ibuprofen, and oral disinfectants (sodium hypochlorite, hypochlorous acid, hydrogen peroxide, among others) for the initial phases of disease progression. On top of these, therapeutic options for patients presenting with pulmonary compromise before or during hospitalization for phase IIb include colchicine, dexamethasone or methylprednisolone, and anticoagulation (rivaroxaban, apixaban, heparin, or enoxaparin).
Period: Overall Study
Arm/Group | Daily Oral Dose of Thymic Peptides | Historic Control Group
Started | 22 | 22
Completed | 20 | 16
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 0 | 5
Not completed — Referred to another hospital before day 20 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Oral Dose of Thymic Peptides | Historic Control Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (16) | 57 (17) | 54 (16)
Age, Customized [Count of Participants; unit: Participants]
  ≤60 years | 15 | 12 | 27
  61-64 years | 2 | 3 | 5
  ≥ 65 years | 5 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 15 | 13 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mestizo | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  Honduras | 22 | 22 | 44
Median no. of days since symptom onset [Median (Inter-Quartile Range); unit: days] | 11.5 [9 to 13] | 10 [9 to 14] | 10.5 [9 to 13]
Comorbidities [Mean (Standard Deviation); unit: Comorbidities] | 2 (1) | 2 (2) | 2 (1)
Coexisting conditions-Diabetes [Count of Participants; unit: Participants] | 11 | 3 | 14
Coexisting conditions-Hypertension [Count of Participants; unit: Participants] | 7 | 9 | 16
Coexisting conditions-Obesity [Count of Participants; unit: Participants] | 2 | 4 | 6
Coexisting conditions-Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 1 | 1 | 2
Coexisting conditions-Heart Failure [Count of Participants; unit: Participants] | 0 | 1 | 1
Coexisting conditions-Organ damage (other than lung) [Count of Participants; unit: Participants] | 12 | 15 | 27
WHO Clinical Progression Score of 5 at hospitalization [Count of Participants; unit: Participants] — WHO Clinical Progression Scale: 0, uninfected; 1, asymptomatic, viral RNA detected; 2, symptomatic and independent; 3, symptomatic and assistance needed; 4, hospitalised, no oxygen therapy; 5, hospitalised, oxygen by mask or nasal prongs; 6, hospitalised, oxygen by non-invasive ventilation or high flow; 7, intubation and mechanical ventilation pO2/FiO2 ≥150 or SpO2/FiO2 ≥200; 8, mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or vasopressors; 9, mechanical ventilation, pO2/FiO2 <150 and vasopressors, dialysis, or ECMO (extracorporeal membrane oxygenation); 10, dead.
  Participants | 22 | 22 | 44
Heart rate distribution [Count of Participants; unit: Participants]
  51-90 beats/min | 14 | 10 | 24
  91-110 beats/min | 6 | 10 | 16
  111-130 beats/min | 2 | 2 | 4
Systolic blood pressure distribution 90-219 mmHg [Count of Participants; unit: Participants] | 22 | 22 | 44
Respiratory rate distribution [Count of Participants; unit: Participants]
  21-24 breaths/min | 2 | 3 | 5
  ≥ 25 breaths/min | 20 | 19 | 39
Oxygen saturation distribution [Count of Participants; unit: Participants]
  92-93% | 3 | 3 | 6
  ≤91% | 19 | 19 | 38
Temperature distribution [Count of Participants; unit: Participants]
  35.6-37.9 °C | 19 | 19 | 38
  38-39 °C | 3 | 2 | 5
  ≥39.1 °C | 0 | 1 | 1
SARS-CoV-2 positive test result [Count of Participants; unit: Participants] | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Time to Participant Recovery
Description: Measured in days to clinical recovery that will be defined as the first day, during the 20 days after enrollment, on which a patient met the criteria for category 1, 2, or 3 on the eight-category ordinal scale. The categories are as follows: 1, not hospitalized and no limitations of activities; 2, not hospitalized, with limitation of activities, home oxygen requirement, or both; 3, hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care; 4, hospitalized, not requiring supplemental oxygen but requiring ongoing medical care (related to Covid-19 or to other medical conditions); 5, hospitalized, requiring any supplemental oxygen; 6, hospitalized, requiring noninvasive ventilation or use of high-flow oxygen devices; 7, hospitalized, receiving invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); and 8, death.
Time Frame: During hospitalization for up to 20 days.
Population: Analyses were performed according to the intention-to-treat principle.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Daily Oral Dose of Thymic Peptides | Historic Control Group
Number analyzed (Participants) | 22 | 22
days | 6 [3.981 to 8.019] | 12 [9.023 to 14.977]

2. Primary Outcome: Number of Participants With Treatment Related Adverse Events as Assessed by the Common Terminology Criteria for Adverse Events Version 5.0
Description: Number of participants who experience adverse events ≥ Grade 3, as defined by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).
Time Frame: Up to 20 days
Population: Only Treatment Related Adverse Event data related to mortality was collected from the Historic Control population.
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Oral Dose of Thymic Peptides | Historic Control Group
Number analyzed (Participants) | 22 | 22
Participants | 0 | 5

3. Primary Outcome: Number of Participants With Treatment Related Side Effects as Assessed by the General Assessment of Side Effects
Description: Number of participants who experience severe side effects as defined by the General Assessment of Side Effects (GASE).
Time Frame: Up to 20 days
Population: Treatment Related Side Effects data not collected from the Historic Control population.
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Oral Dose of Thymic Peptides
Number analyzed (Participants) | 22
Participants | 0

4. Secondary Outcome: Number of Participants That Died by Day 20
Description: Number of participants that died due to any reason by day 20.
Time Frame: Up to 20 days
Population: The analysis assessed the number of patients that died in each arm by day 20.
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Oral Dose of Thymic Peptides | Historic Control Group
Number analyzed (Participants) | 22 | 22
Participants | 0 | 5

ADVERSE EVENTS:
Time Frame: Patients were evaluated daily during their hospitalization, from day 1 through 20. Patients who agreed to follow-ups by phone communication were monitored for adverse events or side effects up to two weeks after discharge.
Description: Adverse events ≥ Grade 3, as defined by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0), were analyzed.
  Only Treatment Related Adverse Event data related to mortality was collected from the Historic Control population.
Arm/Group | Daily Oral Dose of Thymic Peptides | Historic Control Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 5/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 5/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Oral Dose of Thymic Peptides (N=22) | Historic Control Group (N=22)
Death due to respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)

LIMITATIONS AND CAVEATS:
Limitations of this study include its small sample size and the lack of a prospectively randomized control group. This was a single-center study that included only mestizo population, which might have impacted its universal validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT04771013/Prot_SAP_000.pdf